CLINICAL TRIAL: NCT03103256
Title: A Multi-center, Randomized, Double-blind, Parallel-group Phase III Clinical Trial to Evaluate the Efficacy and Safety of YHP1701 Fixed Dose Combination in Patients With Dyslipidemia and Hypertension
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of YHP1701
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YHP1701-301
Record Dates: First submitted 2017-03-22; First posted 2017-04-06 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Hypertension and Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- YHP1701 (Experimental): PO, Once daily (QD), 8 weeks
  Interventions: Drug: YHP1701
- YHR1703 (Active Comparator): PO, Once daily (QD), 8 weeks
  Interventions: Drug: YHR1703
- YHR1704 (Active Comparator): PO, Once daily (QD), 8 weeks
  Interventions: Drug: YHR1704

INTERVENTIONS:
Drug: YHP1701 — PO, Once daily (QD), 8 weeks
  Arms: YHP1701
Drug: YHR1703 — PO, Once daily (QD), 8 weeks
  Arms: YHR1703
Drug: YHR1704 — PO, Once daily (QD), 8 weeks
  Arms: YHR1704

SUMMARY:
The purpose of this study is to determine superiority of YHP1701 comparing to each monotherapy in patient with hypertension and primary hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Both man and woman who is over 19 years old
* Patient with dyslipidemia and hypertension

Exclusion Criteria:

* sSBP difference is ≥20 mmHg or sDBP difference is ≥10 mmHg
* A history of cardiovascular disease
* Rhabdomyolysis, myopathy
* Hypertension or hypercholesterolemia due to secondary causes
* Uncontrolled diabetes
* Evidence of hepatic or renal disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Percent change of LDL-Cholesterol | 0, 8 weeks
  LDL-Cholesterol
Change of mean seated Systolic Blood Pressure | 0, 8 weeks
  Blood Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lee, Study Director — Yuhan Corporation
Locations (1):
- Seoul Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim W, Chang K, Cho EJ, Ahn JC, Yu CW, Cho KI, Kim YJ, Kang DH, Kim SY, Lee SH, Kim U, Kim SJ, Ahn YK, Lee CH, Shin JH, Kim M, Park CG. A randomized, double-blind clinical trial to evaluate the efficacy and safety of a fixed-dose combination of amlodipine/rosuvastatin in patients with dyslipidemia and hypertension. J Clin Hypertens (Greenwich). 2020 Feb;22(2):261-269. doi: 10.1111/jch.13774. Epub 2020 Jan 31. PMID 32003938